CLINICAL TRIAL: NCT02513732
Title: XIENCE Xpedition Everolimus-Eluting Coronary Stent Japan Post Marketing Surveillance
Brief Title: XIENCE Xpedition Everolimus-Eluting Coronary Stent Japan Post Marketing Surveillance (XIENCE Xpedition SV Japan PMS)
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-306
Record Dates: First submitted 2015-07-17; First posted 2015-08-03 (Estimated); Results first posted 2019-02-21 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Ischemic Heart Disease; Angina Pectoris; Coronary Artery Disease; Myocardial Ischemia
Keywords: Drug Eluting Stent; Coronary Stent; Everolimus; Stent Thrombosis
MeSH Terms: conditions — Myocardial Ischemia; Angina Pectoris; Coronary Artery Disease | interventions — Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- XIENCE Xpedition 2.25 mm stent arm: Patients receiving XIENCE Xpedition 2.25 mm stent
  Interventions: Device: XIENCE Xpedition 2.25 mm stent

INTERVENTIONS:
Device: XIENCE Xpedition 2.25 mm stent — Patients receiving XIENCE Xpedition 2.25 mm stent

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of XIENCE Xpedition Everolimus-Eluting 2.25mm Stent in real world practice in Japanese hospitals.

DETAILED DESCRIPTION:
Based on Good Post-marketing Study Practice (GPSP) regulation, general patient population with ischemic heart disease who are eligible for treatment with XIENCE Xpedition Everolimus-Eluting 2.25mm Stent will be registered, with no particular inclusion/exclusion criteria, and may be eligible for angiographic follow-up at eight months and clinical follow-up at one year.

The XIENCE Xpedition 2.25 mm stent is composed of the stent identical to the stent of the XIENCE PRIME SV Stent.Therefore, the data collected from the PMS will be pooled with data collected from the ongoing XIENCE PRIME SV PMS for analysis.

ELIGIBILITY:
1. Inclusion criteria

   1. Patient informed consent is required for registration of this PMS. In cases where patient informed consent (or providing some type of information) is required for PMS per the participating site policy, the Sponsor will cooperate as needed.
   2. Patients who are treated by XIENCE Xpedition 2.25mm stent will be registered.

      * The observations will be compiled on a per-patient basis even if multiple XIENCE Xpedition 2.25mm stents are implanted during the index procedure.
      * A patient whose side-branch is treated by XIENCE Xpedition 2.25mm stent can be registered. In such a case, main vessel should be treated by XIENCE Xpedition.
      * The observations will not be compiled on a per-patient basis if a patient is treated by XIENCE Xpedition 2.25mm stent overlapped with other stents for bail-out purpose.
      * Additional revascularization procedures as a part of adverse event treatment and planned staged procedures will not be considered as another registration, or adverse events.
      * A patient who is treated, but failed to be implanted by XIENCE Xpedition 2.25mm stent and finally treated by other devices only (No XIENCE Xpedition 2.25mm stent are implanted) must also be registered. In such a case, only the stent information, device deficiency information and reportable adverse events related to the Xpedition stent, if any, are required to be captured. Follow-up of the patient who does not receive any XIENCE Xpedition 2.25mm stent is not required.
2. Exclusion criteria

   1. If it is known at the time of index procedure that the patient is not able to return for the 8-month follow-up visit for angiogram and for the 1-year clinical follow-up, then the patient should not be registered in the PMS.
   2. Patients who are attending or will attend other PMS with invasive medical procedure will not be registered.
3. A patient may have another lesion(s) that may be treated by larger diameter (≥ 2.5mm) stent(s). In such a case, treatment by XIENCE Xpedition is preferable. Lesion(s) treated by other than XIENCE Xpedition 2.25mm stent is not considered as the target lesion.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General patient population with ischemic heart disease in Japan who are eligible for treatment with XIENCE Xpedition 2.25 mm stent will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-07; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Kozuma, MD, Study Chair — Teikyo University Hospital, Tokyo
Locations (11):
- Japan (11):
  - Hyogo Prefectural Amagasaki Hospital, Hyōgo
  - Ishikawa Prefectural Central Hospital, Ishikawa
  - Miyazaki Medical Association Hospital, Miyazaki
  - Osaka Police Hospital, Osaka
  - Hanaoka Seishu Memorial Cardiovascular Clinic, Sapporo
  - JCHO Hokkaido Hospital, Sapporo
  - Tokushima Red Cross Hospital, Tokushima
  - Mitsui Memorial Hospital, Tokyo
  - Toranomon Hospital, Tokyo
  - Teikyo University Hospital, Tokyo
  - Showa University Fujigaoka Hospital, Yokohama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 100 subjects were enrolled from multiple sites.
Period: Overall Study
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Started | 100
Completed | 78
Not Completed | 22
Not completed — Lost to Follow-up | 11
Not completed — Death | 9
Not completed — Changing hospital | 2

BASELINE CHARACTERISTICS:
Population: A total of 100 patients were treated with Xience Xpedition 2.25 mm stent
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 100
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 100
Region of Enrollment [Number; unit: participants]
  Japan | 100
Height [Mean (Standard Deviation); unit: cm] | 162.58 (8.31)
Weight [Mean (Standard Deviation); unit: kg] | 64.22 (10.05)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.23 (2.82)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stent Thrombosis: Late
Description: Scaffold/Stent thrombosis should be reported as a cumulative value at the different time points and with the different separate time points. Time 0 is defined as the time point after the guiding catheter has been removed and the subject left the catheterization lab.
  Timings:
  Acute scaffold/stent thrombosis : 0 - 24 hours post stent implantation Subacute scaffold/stent thrombosis: >24 hours - 30 days post stent implantation Late scaffold/stent thrombosis: 30 days - 1 year post stent implantation Very late scaffold/stent thrombosis: >1 year post stent implantation
Time Frame: 30 days to 1 year post stent implantation-Day 212
Population: Intend To Treat population(ITT population)
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 1

2. Secondary Outcome: Percent Diameter Stenosis (%DS)
Description: In-segment, In-stent, Proximal and Distal. The value calculated as 100 * (1 - minimum lumen diameter/reference vessel diameter) (MLD/RVD) using the mean values from two orthogonal views (when possible) by quantitative coronary angiography (QCA).
Time Frame: Pre-procedure
Population: ITT population
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Units Other Than Participants: Number of lesions
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Number analyzed (Number of lesions) | 120
Percent Diameter stenosis | 72.02 (16.97)

3. Secondary Outcome: Percent Diameter Stenosis (%DS)
Description: In-segment, In-stent, Proximal and Distal. The value calculated as 100 * (1 - MLD/RVD) using the mean values from two orthogonal views (when possible) by quantitative coronary angiography (QCA).
Time Frame: Immediately after the procedure
Population: ITT population
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Units Other Than Participants: Number of lesions
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Number analyzed (Number of lesions) | 120
Percent Diameter stenosis | 23.15 (12.01)

4. Secondary Outcome: Percent Diameter Stenosis (%DS)
Description: as for outcome 3
Time Frame: During follow-up, at 8 months post procedure
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: Percent Diameter Stenosis
Units Other Than Participants: Number of lesions
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 77
Number analyzed (Number of lesions) | 79
Percent Diameter Stenosis | 32.14 (20.43)

5. Secondary Outcome: Number of Participants Using Antiplatelet Therapy
Description: Number of patients using aspirin, clopidogrel, ticlopidine, cilostazol,prasugrel, compounding agents and other agents.
Time Frame: At baseline before procedure
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants
  Aspirin + clopidogrel | 68
  Aspirin + ticlopidine | 2
  Aspirin | 92
  Clopidogrel | 67
  Ticlodipine | 2
  Cilostazol | 3
  Prasugrel | 25
  Compounding agent | 6
  Other | 2

6. Secondary Outcome: Number of Participants Using Antiplatelet Therapy
Description: Number of patients using aspirin, clopidogrel, ticlopidine, cilostazol,prasugrel, compounding agents and other agents.
Time Frame: Date of discharge from procedure day
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants
  Aspirin + clopidogrel | 62
  Aspirin + ticlopidine | 2
  Aspirin | 79
  Clopidogrel | 61
  Ticlodipine | 2
  Cilostazol | 2
  Prasugrel | 17
  Compounding agent | 6
  Other | 2

7. Secondary Outcome: Number of Participants Using Antiplatelet Therapy
Description: Number of patients using aspirin, clopidogrel, ticlopidine, cilostazol,prasugrel, compounding agents and other agents.
Time Frame: 8 months observation day from the procedure day
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants
  Aspirin + clopidogrel | 54
  Aspirin + ticlopidine | 2
  Aspirin | 70
  Clopidogrel | 52
  Ticlodipine | 2
  Cilostazol | 2
  Prasugrel | 7
  Compounding agent | 5
  Other | 1

8. Secondary Outcome: Number of Participants Using Antiplatelet Therapy
Description: Number of patients using aspirin, clopidogrel, ticlopidine, cilostazol,prasugrel, compounding agents and other agents.
Time Frame: 1 year observation day from the procedure day
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 98
Participants
  Aspirin + clopidogrel | 43
  Aspirin + ticlopidine | 1
  Aspirin | 67
  Clopidogrel | 44
  Ticlodipine | 1
  Cilostazol | 2
  Prasugrel | 6
  Compounding agent | 4
  Other | 1

9. Secondary Outcome: Number of Participants Using Antiplatelet Therapy
Description: Number of patients using aspirin, clopidogrel, ticlopidine, cilostazol,prasugrel, compounding agents and other agents.
Time Frame: 2 years observation day from the procedure day
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 96
Participants
  Aspirin + clopidogrel | 31
  Aspirin + ticlopidine | 1
  Aspirin | 64
  Clopidogrel | 33
  Ticlodipine | 1
  Cilostazol | 2
  Prasugrel | 4
  Compounding agent | 4
  Other | 1

10. Secondary Outcome: Number of Participants Using Antiplatelet Therapy
Description: Number of patients using aspirin, clopidogrel, ticlopidine, cilostazol,prasugrel, compounding agents and other agents.
Time Frame: 3 years observation day from the procedure day
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 95
Participants
  Aspirin + clopidogrel | 29
  Aspirin + ticlopidine | 1
  Aspirin | 60
  Clopidogrel | 31
  Ticlodipine | 1
  Cilostazol | 2
  Prasugrel | 4
  Compounding agent | 4
  Other | 1

11. Secondary Outcome: Number of Participants Using Antiplatelet Therapy
Description: Number of patients using aspirin, clopidogrel, ticlopidine, cilostazol,prasugrel, compounding agents and other agents.
Time Frame: 4 years observation day from the procedure day
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 94
Participants
  Aspirin + clopidogrel | 26
  Aspirin + ticlopidine | 1
  Aspirin | 59
  Clopidogrel | 27
  Prasugrel | 3
  Ticlodipine | 1
  Cilostazol | 2
  Compounding agent | 4
  Other | 1

12. Secondary Outcome: Number of Participants Using Antiplatelet Therapy
Description: Number of patients using aspirin, clopidogrel, ticlopidine, cilostazol,prasugrel, compounding agents and other agents.
Time Frame: 5 years observation day from the procedure day
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 91
Participants
  Aspirin + clopidogrel | 23
  Aspirin + ticlopidine | 1
  Aspirin | 52
  Clopidogrel | 23
  Prasugrel | 4
  Ticlodipine | 1
  Cilostazol | 2
  Compounding agent | 3
  Other | 1

13. Secondary Outcome: Number of Participants With Death
Description: All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Specifically, any unexpected death even in subjects with coexisting potentially fatal non-cardiac disease (e.g. cancer, infection) should be classified as cardiac.
  * Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  * Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  * Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
Time Frame: During hospitalization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

14. Secondary Outcome: Number of Participants With Death
Description: as for outcome 13
Time Frame: 0 to 8 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

15. Secondary Outcome: Number of Participants With Death
Description: as for outcome 13
Time Frame: 0 to 1 year
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 1

16. Secondary Outcome: Number of Participants With Death
Description: as for outcome 13
Time Frame: 0 to 2 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 4

17. Secondary Outcome: Number of Participants With Death
Description: as for outcome 13
Time Frame: 0 to 3 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 7

18. Secondary Outcome: Number of Participants With Death
Description: as for outcome 13
Time Frame: 0 to 4 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 8

19. Secondary Outcome: Number of Participants With Death
Description: as for outcome 13
Time Frame: 0 to 5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 9

20. Secondary Outcome: Number of Participants With Target Lesion Revascularization Based on Ischemia Findings
Description: Target lesion revascularization is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion.
Time Frame: During hospitalization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

21. Secondary Outcome: Number of Participants With Target Lesion Revascularization Based on Ischemia Findings
Description: as for outcome 20
Time Frame: 0 to 8 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 1

22. Secondary Outcome: Number of Participants With Target Lesion Revascularization Based on Ischemia Findings
Description: as for outcome 20
Time Frame: 0 to 1 year
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 3

23. Secondary Outcome: Number of Participants With Target Lesion Revascularization Based on Ischemia Findings
Description: as for outcome 20
Time Frame: 0 to 2 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 4

24. Secondary Outcome: Number of Participants With Target Lesion Revascularization Based on Ischemia Findings
Description: as for outcome 20
Time Frame: 0 to 3 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 6

25. Secondary Outcome: Number of Participants With Target Lesion Revascularization Based on Ischemia Findings
Description: as for outcome 20
Time Frame: 0 to 4 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 6

26. Secondary Outcome: Number of Participants With Target Lesion Revascularization Based on Ischemia Findings
Description: as for outcome 20
Time Frame: 0 to 5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 6

27. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: Myocardial Infarction (MI) - Q wave MI: Development of new, pathological Q wave on the ECG.
  -Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: During hospitalization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

28. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: as for outcome 27
Time Frame: 0 to 8 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

29. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: as for outcome 27
Time Frame: 0 to 1 year
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 1

30. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: as for outcome 27
Time Frame: 0 to 2 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 1

31. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: as for outcome 27
Time Frame: 0 to 3 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 1

32. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: as for outcome 27
Time Frame: 0 to 4 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 1

33. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: as for outcome 27
Time Frame: 0 to 5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 1

34. Secondary Outcome: Number of Participants With Cardiac Death
Description: Cardiac death is defined as any death in which a cardiac cause cannot be excluded. (This includes but is not limited to acute myocardial infarction, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality,cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery.)
Time Frame: During hospitalization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

35. Secondary Outcome: Number of Participants With Cardiac Death
Description: as for outcome 34
Time Frame: 0 to 8 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

36. Secondary Outcome: Number of Participants With Cardiac Death
Description: as for outcome 34
Time Frame: 0 to 1 year
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

37. Secondary Outcome: Number of Participants With Cardiac Death
Description: as for outcome 34
Time Frame: 0 to 2 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

38. Secondary Outcome: Number of Participants With Cardiac Death
Description: as for outcome 34
Time Frame: 0 to 3 Years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

39. Secondary Outcome: Number of Participants With Cardiac Death
Description: as for outcome 34
Time Frame: 0 to 4 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

40. Secondary Outcome: Number of Participants With Cardiac Death
Description: as for outcome 34
Time Frame: 0 to 5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

41. Secondary Outcome: Number of Participants With MI Related to Target Vessel
Description: as for outcome 27
Time Frame: During hospitalization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

42. Secondary Outcome: Number of Participants With MI Related to Target Vessel
Description: as for outcome 27
Time Frame: 0 to 8 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

43. Secondary Outcome: Number of Participants With MI Related to Target Vessel
Description: as for outcome 27
Time Frame: 0 to 1 year
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

44. Secondary Outcome: Number of Participants With MI Related to Target Vessel
Description: as for outcome 27
Time Frame: 0 to 2 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

45. Secondary Outcome: Number of Participants With MI Related to Target Vessel
Description: as for outcome 27
Time Frame: 0 to 3 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

46. Secondary Outcome: Number of Participants With MI Related to Target Vessel
Description: as for outcome 27
Time Frame: 0 to 4 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

47. Secondary Outcome: Number of Participants With MI Related to Target Vessel
Description: as for outcome 27
Time Frame: 0 to 5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

48. Secondary Outcome: Number of Participants With Death,Myocardial Infarction and Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: During hospitalization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 2

49. Secondary Outcome: Number of Participants With Death,Myocardial Infarction and Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: 0 to 8 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 23

50. Secondary Outcome: Number of Participants With Death,Myocardial Infarction and Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: 0 to 1 year
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 29

51. Secondary Outcome: Number of Participants With Death,Myocardial Infarction and Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: 0 to 2 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 41

52. Secondary Outcome: Number of Participants With Death,Myocardial Infarction and Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: 0 to 3 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 47

53. Secondary Outcome: Number of Participants With Death,Myocardial Infarction and Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: 0 to 4 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 48

54. Secondary Outcome: Number of Participants With Death,Myocardial Infarction and Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: 0 to 5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 50

55. Secondary Outcome: Number of Participants With All Revascularization
Description: All revascularization endpoint is comprised of TLR, TVR excluding TLR, and non-TVR.
Time Frame: During hospitalization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 2

56. Secondary Outcome: Number of Participants With All Revascularization
Description: All revascularization endpoint is comprised of TLR, TVR excluding TLR, and non-TVR.
Time Frame: 0 to 8 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 23

57. Secondary Outcome: Number of Participants With All Revascularization
Description: All revascularization endpoint is comprised of TLR, TVR excluding TLR, and non-TVR.
Time Frame: 0 to 1 year
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 29

58. Secondary Outcome: Number of Participants With All Revascularization
Description: All revascularization endpoint is comprised of TLR, TVR excluding TLR, and non-TVR.
Time Frame: 0 to 2 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 38

59. Secondary Outcome: Number of Participants With All Revascularization
Description: All revascularization endpoint is comprised of TLR, TVR excluding TLR, and non-TVR.
Time Frame: 0 to 3 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 41

60. Secondary Outcome: Number of Participants With All Revascularization
Description: All revascularization endpoint is comprised of TLR, TVR excluding TLR, and non-TVR.
Time Frame: 0 to 4 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 42

61. Secondary Outcome: Number of Participants With All Revascularization
Description: All revascularization endpoint is comprised of TLR, TVR excluding TLR, and non-TVR.
Time Frame: 0 to 5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 44

62. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: Target Vessel Failure (TVF) is the composite of Cardiac Death, Myocardial infarction (MI) or Ischemic-Driven Target Vessel Revascularization (ID-TVR).
Time Frame: During hospitalization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

63. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 62
Time Frame: 0 to 8 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 2

64. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 62
Time Frame: 0 to 1 year
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 6

65. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 62
Time Frame: 0 to 2 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 7

66. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 62
Time Frame: 0 to 3 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 9

67. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 62
Time Frame: 0 to 4 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 10

68. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 62
Time Frame: 0 to 5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 11

69. Secondary Outcome: Number of Participants With Target Vessel Revascularization (Non-TLR)
Description: Target vessel revascularization (TVR) includes ischemia driven TVR, non-TLR and non- ischemia driven TVR, non-TLR.
Time Frame: During hospitalization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 2

70. Secondary Outcome: Number of Participants With Target Vessel Revascularization (Non-TLR)
Description: Target vessel revascularization (TVR) includes ischemia driven TVR, non-TLR and non- ischemia driven TVR, non-TLR.
Time Frame: 0 to 8 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 6

71. Secondary Outcome: Number of Participants With Target Vessel Revascularization (Non-TLR)
Description: Target vessel revascularization (TVR) includes ischemia driven TVR, non-TLR and non- ischemia driven TVR, non-TLR.
Time Frame: 0 to 1 year
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 7

72. Secondary Outcome: Number of Participants With Target Vessel Revascularization (Non-TLR)
Description: Target vessel revascularization (TVR) includes ischemia driven TVR, non-TLR and non- ischemia driven TVR, non-TLR.
Time Frame: 0 to 2 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 9

73. Secondary Outcome: Number of Participants With Target Vessel Revascularization (Non-TLR)
Description: Target vessel revascularization (TVR) includes ischemia driven TVR, non-TLR and non- ischemia driven TVR, non-TLR.
Time Frame: 0 to 3 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 11

74. Secondary Outcome: Number of Participants With Target Vessel Revascularization (Non-TLR)
Description: Target vessel revascularization (TVR) includes ischemia driven TVR, non-TLR and non- ischemia driven TVR, non-TLR.
Time Frame: 0 to 4 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 12

75. Secondary Outcome: Number of Participants With Target Vessel Revascularization (Non-TLR)
Description: Target vessel revascularization (TVR) includes ischemia driven TVR, non-TLR and non- ischemia driven TVR, non-TLR.
Time Frame: 0 to 5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 13

76. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TLR or TVR (Non-TLR))
Description: Target vessel revascularization (TLR or TVR, non-TLR) includes ischemia driven TVR (TLR or TVR, non-TLR) or non-ischemia driven TVR (TLR or TVR, nonTLR).
Time Frame: During hospitalization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 2

77. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TLR or TVR (Non-TLR))
Description: as for outcome 76
Time Frame: 0 to 8 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 11

78. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TLR or TVR (Non-TLR))
Description: as for outcome 76
Time Frame: 0 to 1 year
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 16

79. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TLR or TVR (Non-TLR))
Description: as for outcome 76
Time Frame: 0 to 2 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 19

80. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TLR or TVR (Non-TLR))
Description: as for outcome 76
Time Frame: 0 to 3 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 22

81. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TLR or TVR (Non-TLR))
Description: as for outcome 76
Time Frame: 0 to 4 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 23

82. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TLR or TVR (Non-TLR))
Description: as for outcome 76
Time Frame: 0 to 5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 24

83. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TLR (Major Adverse Cardiac Events-MACE)
Description: Major adverse cardiac events (MACE) is defined as the composite of cardiac death, all myocardial infarction, and ischemic driven target lesion revascularization (ID-TLR).
Time Frame: During hospitalization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

84. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TLR (Major Adverse Cardiac Events-MACE)
Description: as for outcome 83
Time Frame: 0 to 8 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 1

85. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TLR (Major Adverse Cardiac Events-MACE)
Description: as for outcome 83
Time Frame: 0 to 1 year
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 4

86. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TLR (Major Adverse Cardiac Events-MACE)
Description: as for outcome 83
Time Frame: 0 to 2 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 5

87. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TLR (Major Adverse Cardiac Events-MACE)
Description: as for outcome 83
Time Frame: 0 to 3 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 7

88. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TLR (Major Adverse Cardiac Events-MACE)
Description: as for outcome 83
Time Frame: 0 to 4 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 8

89. Secondary Outcome: Number of Participants With Cardiac Death/All MI/ID-TLR (Major Adverse Cardiac Events-MACE)
Description: as for outcome 83
Time Frame: 0 to 5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 8

90. Secondary Outcome: Number of Participants With Death/All MI
Description: All deaths includes Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
  Myocardial Infarction (MI) - Q wave MI: Development of new, pathological Q wave on the ECG.
  -Non-Q wave MI: Those MIs which are not Q-wave MI
Time Frame: During hospitalization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

91. Secondary Outcome: Number of Participants With Death/All MI
Description: as for outcome 90
Time Frame: 0 to 8 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

92. Secondary Outcome: Number of Participants With Death/All MI
Description: as for outcome 90
Time Frame: 0 to 1 year
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 2

93. Secondary Outcome: Number of Participants With Death/All MI
Description: as for outcome 90
Time Frame: 0 to 2 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 5

94. Secondary Outcome: Number of Participants With Death/All MI
Description: as for outcome 90
Time Frame: 0 to 3 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 8

95. Secondary Outcome: Number of Participants With Death/All MI
Description: as for outcome 90
Time Frame: 0 to 4 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 10

96. Secondary Outcome: Number of Participants With Death/All MI
Description: as for outcome 90
Time Frame: 0 to 5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 11

97. Secondary Outcome: Number of Participants With Cardiac Death/All MI
Description: as for outcome 90
Time Frame: During hospitalization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

98. Secondary Outcome: Number of Participants With Cardiac Death/All MI
Description: as for outcome 90
Time Frame: 0 to 8 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

99. Secondary Outcome: Number of Participants With Cardiac Death/All MI
Description: as for outcome 90
Time Frame: 0 to 1 year
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 1

100. Secondary Outcome: Number of Participants With Cardiac Death/All MI
Description: as for outcome 90
Time Frame: 0 to 2 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 1

101. Secondary Outcome: Number of Participants With Cardiac Death/All MI
Description: as for outcome 90
Time Frame: 0 to 3 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 1

102. Secondary Outcome: Number of Participants With Cardiac Death/All MI
Description: as for outcome 90
Time Frame: 0 to 4 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 2

103. Secondary Outcome: Number of Participants With Cardiac Death/All MI
Description: as for outcome 90
Time Frame: 0 to 5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 2

104. Secondary Outcome: Number of Participants With Cardiac Death or Target-Vessel MI
Description: Cardiac death is defined as any death in which a cardiac cause cannot be excluded. (This includes but is not limited to acute myocardial infarction, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality,cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery).
Time Frame: During hospitalization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

105. Secondary Outcome: Number of Participants With Cardiac Death or Target-Vessel MI
Description: as for outcome 104
Time Frame: 0 to 8 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

106. Secondary Outcome: Number of Participants With Cardiac Death or Target-Vessel MI
Description: as for outcome 104
Time Frame: 0 to 1 year
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

107. Secondary Outcome: Number of Participants With Cardiac Death or Target-Vessel MI
Description: as for outcome 104
Time Frame: 0 to 2 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

108. Secondary Outcome: Number of Participants With Cardiac Death or Target-Vessel MI
Description: as for outcome 104
Time Frame: 0 to 3 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

109. Secondary Outcome: Number of Participants With Cardiac Death or Target-Vessel MI
Description: as for outcome 104
Time Frame: 0 to 4 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

110. Secondary Outcome: Number of Participants With Cardiac Death or Target-Vessel MI
Description: as for outcome 104
Time Frame: 0 to 5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

111. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: TLF is defined as composite of Cardiac Death, Myocardial Infarction (per protocol-defined MI definition), attributable to Target Vessel (TV-MI), or Ischemic-Driven Target Lesion Revascularization (ID-TLR).
Time Frame: During hospitalization
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 0

112. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: as for outcome 111
Time Frame: 0 to 8 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 1

113. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: as for outcome 111
Time Frame: 0 to 1 year
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 3

114. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: as for outcome 111
Time Frame: 0 to 2 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 4

115. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: as for outcome 111
Time Frame: 0 to 3 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 6

116. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: as for outcome 111
Time Frame: 0 to 4 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 6

117. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: as for outcome 111
Time Frame: 0 to 5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Participants | 6

118. Secondary Outcome: Mean Acute Gain: In-stent, In-segment
Description: The difference between post- and pre-procedural MLD.
Time Frame: At 8 months, post index procedure
Population: ITT population
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Number of lesions QCA
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Number analyzed (Number of lesions QCA) | 120
mm
  Stent | 1.51 (0.46)
  Segment | 1.20 (0.50)

119. Secondary Outcome: Mean Late Loss(LL): In-stent, In-segment, Proximal, and Distal
Description: Late loss is calculated as MLD post procedure - MLD at follow-up.
Time Frame: At 8 months, post index procedure
Population: ITT population
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Number of lesions QCA
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Number analyzed (Number of lesions QCA) | 120
mm
  Stent | 0.28 (0.36)
  Proximal | 0.03 (0.36)
  Distal | -0.06 (0.28)
  Segment | 0.20 (0.50)

120. Secondary Outcome: Mean Net Gain: In-stent, In-segment
Description: Late procedural outcome is influenced by both the acute gain provided by the intervention (pre to post) and the subsequent late loss that occurs after the intervention (post to follow-up).The net gain is thus the sum of the offsetting effects of acute gain and late loss (net gain = acute gain - late loss).
Time Frame: At 8 months, post index procedure
Population: ITT population
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Number of lesions QCA
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Number analyzed (Number of lesions QCA) | 120
mm
  Stent | 1.26 (0.52)
  Segment | 1.04 (0.62)

121. Secondary Outcome: Mean Lesion Length
Description: The lesion length will be measured by QCA.
Time Frame: Pre-procedure
Population: ITT population
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Number of lesions QCA
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Number analyzed (Number of lesions QCA) | 120
mm | 17.38 (10.27)

122. Secondary Outcome: Minimum Blood Vessel Diameter
Description: Minimum blood vessel diameter measured by QCA
Time Frame: Pre-procedure
Population: ITT population
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Number of lesions QCA
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Number analyzed (Number of lesions QCA) | 120
mm | 0.55 (0.34)

123. Secondary Outcome: Minimum Blood Vessel Diameter
Description: Minimum blood vessel diameter measured by QCA
Time Frame: Immediately after the procedure
Population: ITT population
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Number of lesions QCA
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Number analyzed (Number of lesions QCA) | 120
mm | 2.03 (0.27)

124. Secondary Outcome: Minimum Blood Vessel Diameter
Description: Minimum blood vessel diameter measured by QCA
Time Frame: During follow-up, at 8 months post procedure
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Number of lesions QCA
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 77
Number analyzed (Number of lesions QCA) | 79
mm | 1.54 (0.51)

125. Secondary Outcome: Mean Reference Vessel Diameter (RVD)
Description: Reference vessel diameter measured by QCA
Time Frame: Pre-procedure
Population: ITT population.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Number of lesions
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Number analyzed (Number of lesions) | 120
mm | 2.04 (0.36)

126. Secondary Outcome: Mean Reference Vessel Diameter (RVD)
Description: Reference vessel diameter measured by QCA
Time Frame: Immediately after the procedure
Population: ITT population.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Number of lesions QCA
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 100
Number analyzed (Number of lesions QCA) | 120
mm | 2.34 (0.37)

127. Secondary Outcome: Mean Reference Vessel Diameter (RVD)
Description: Reference vessel diameter measured by QCA
Time Frame: During follow-up, at 8 months post procedure
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Number of lesions QCA
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
Number analyzed (Participants) | 77
Number analyzed (Number of lesions QCA) | 79
mm | 2.28 (0.38)

ADVERSE EVENTS:
Time Frame: 5 Years
Description: In this surveillance, Investigators report Serious Adverse event, Cardiac Adverse Event, DAPT related AE and Device Deficiency as per local regulation and protocol.
Arm/Group | XIENCE Xpedition 2.25 mm Stent Arm
All-Cause Mortality (participants affected / at risk) | 9/100
Serious Adverse Events (participants affected / at risk) | 63/100
Other Adverse Events (participants affected / at risk) | 67/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XIENCE Xpedition 2.25 mm Stent Arm (N=100)
Bacteraemia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Pyelonephritis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Infectious peritonitis (Infections and infestations) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Contrast media allergy (Immune system disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Cervical myelopathy (Nervous system disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 12
Angina unstable (Cardiac disorders) | 3
Cardiac failure (Cardiac disorders) | 4
Coronary artery stenosis (Cardiac disorders) | 23
Ventricular tachycardia (Cardiac disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Peripheral artery aneurysm (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 7
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 7
Colonic polyp (Gastrointestinal disorders) | 2
Enteritis (Gastrointestinal disorders) | 1
Gastric ulcer hemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatic mass (Hepatobiliary disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Asthenia (General disorders) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral hemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 2
Cardiac failure chronic (Cardiac disorders) | 2
Prinzmetal angina (Cardiac disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 1
Hematochezia (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Nephropathy toxic (Renal and urinary disorders) | 1
Bladder tamponade (Renal and urinary disorders) | 2
Prostatitis (Reproductive system and breast disorders) | 1
Death (General disorders) | 3
Pyrexia (General disorders) | 1
Device-related thrombosis (General disorders) | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 20
Heat illness (Injury, poisoning and procedural complications) | 1
Aortic valve stenosis (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XIENCE Xpedition 2.25 mm Stent Arm (N=100)
Bacteraemia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Pyelonephritis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Infectious peritonitis (Infections and infestations) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Contrast media allergy (Immune system disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Cervical myelopathy (Nervous system disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 15
Angina unstable (Cardiac disorders) | 3
Cardiac failure (Cardiac disorders) | 4
Coronary artery stenosis (Cardiac disorders) | 27
Ventricular tachycardia (Cardiac disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Peripheral artery aneurysm (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 7
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 7
Colonic polyp (Gastrointestinal disorders) | 2
Enteritis (Gastrointestinal disorders) | 1
Gastric ulcer hemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatic mass (Hepatobiliary disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Asthenia (General disorders) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral hemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 2
Cardiac failure chronic (Cardiac disorders) | 2
Prinzmetal angina (Cardiac disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 1
Hematochezia (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Nephropathy toxic (Renal and urinary disorders) | 1
Bladder tamponade (Renal and urinary disorders) | 2
Prostatitis (Reproductive system and breast disorders) | 1
Death (General disorders) | 3
Pyrexia (General disorders) | 1
Device-related thrombosis (General disorders) | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 23
Heat illness (Injury, poisoning and procedural complications) | 1
Aortic valve stenosis (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Retinal hemorrhage (Eye disorders) | 1
Coronary artery dissection (Cardiac disorders) | 1
Coronary artery no-reflow (Cardiac disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2014-05-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT02513732/Prot_000.pdf
  • Statistical Analysis Plan (2015-06-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT02513732/SAP_001.pdf